CLINICAL TRIAL: NCT05924568
Title: Assessment of Strength Outcomes After Use of the PrimusRS for Specificity of Training in a Cardiac Rehabilitation Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brandon Hathorn (Other)
Collaborators: Baylor Heart and Vascular Institute Cardiovascular Research Review Committee (Unknown)
Responsible Party: Sponsor-Investigator, Brandon Hathorn, Clinical Exercise Physiologist, Baylor Research Institute
Organization: Baylor Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Purpose: Treatment
Other Study IDs: 015-050
Record Dates: First submitted 2023-06-21; First posted 2023-06-29 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Coronary Artery Disease; Valve Disease, Heart
Keywords: Coronary artery bypass graft; Valve replacement; Valve Repair; Median Sternotomy
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Median Sternotomy (Experimental)
  Interventions: Other: Educational session with Keep Your Move in the Tube and PrimusRS

INTERVENTIONS:
Other: Educational session with Keep Your Move in the Tube and PrimusRS

SUMMARY:
The purpose of this study is to determine if performed force measurements yield a different recommended weight lifted during the sternotomy healing process than the traditional gold standard of 5 pounds. A secondary endpoint data obtained will be scores from the pre and post-activity questionnaires.

DETAILED DESCRIPTION:
In a prospective study involving 130 cardiac rehabilitation patients muscular strength will be measured with a force dynamometer (PRIMUS) on six commonly performed activities. During the first session of cardiac rehabilitation, each subject's date of birth, height, and weight will be recorded. To ensure safety, cardiovascular nurse specialists and exercise physiologists will monitor the patients for hypertension (blood pressure >240/110 mm Hg), arrhythmias, angina, dizziness, pain, shortness of breath, and perceived exertion. The subjects will be asked to complete a pre-activity confidence survey. On the second day of cardiac rehabilitation, a clinical exercise specialist will the PRIMUS equipment to obtain force measurements on the six activities including: rising from a bed, rising from a chair, opening a door, lifting an object from the floor and/or placing an object overhead. Following the performance of the activities, the patients will be asked to complete a post-activity confidence survey.

ELIGIBILITY:
Inclusion Criteria:

* CABG through median sternotomy
* Valve repair or replacement through median sternotomy
* Any ethic of socio-economic status

Exclusion Criteria:

* Refusal to participate
* Sternal dehiscence
* Permanent pacemaker
* Permanent defibrillator
* Unstable angina
* History of heart transplant
* History of hernia
* History of aneurysm
* Physical disability that limits resistance training
* Uncontrolled hypertension (systolic 160 mmHg or diastolic > 100 mmHg)
* Symptomatic dysrhythmias
* History of aortic dissection

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2015-05-13 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Force pounds lifted post-median sternotomy | Day 1 or 2 of protocol
  Determining if performed force measurements yield a different recommended weight lifted during the sternotomy healing process than the traditional gold standard of 5 pounds.

SECONDARY OUTCOMES:
Changes in confidence to perform ADLs | Day 1 or 2 of protocol
  Change in confidence for ADLs post-sternotomy with a questionnaire pre and post protocol (Scale: 1-5; with 1 being the least confident and 5 being the most confident)

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Hathorn, B.S., Principal Investigator — Baylor Scott and White Health Heart and Vascular Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams J, Schmid J, Parker RD, Coast JR, Cheng D, Killian AD, McCray S, Strauss D, McLeroy Dejong S, Berbarie R. Comparison of force exerted on the sternum during a sneeze versus during low-, moderate-, and high-intensity bench press resistance exercise with and without the valsalva maneuver in healthy volunteers. Am J Cardiol. 2014 Mar 15;113(6):1045-8. doi: 10.1016/j.amjcard.2013.11.064. Epub 2013 Dec 25. PMID 24440333
- [Background] Adams J, Cheng D, Lee J, Shock T, Kennedy K, Pate S. Use of the bootstrap method to develop a physical fitness test for public safety officers who serve as both police officers and firefighters. Proc (Bayl Univ Med Cent). 2014 Jul;27(3):199-202. doi: 10.1080/08998280.2014.11929107. PMID 24982558
- [Background] Adams J, DeJong S, Arnett JK, Kennedy K, Franklin JO, Berbarie RF. High-intensity cardiac rehabilitation training of a firefighter after placement of an implantable cardioverter-defibrillator. Proc (Bayl Univ Med Cent). 2014 Jul;27(3):226-8. doi: 10.1080/08998280.2014.11929118. PMID 24982569
- [Background] Adams J, Cheng D, Berbarie RF. High-intensity, occupation-specific training in a series of firefighters during phase II cardiac rehabilitation. Proc (Bayl Univ Med Cent). 2013 Apr;26(2):106-8. doi: 10.1080/08998280.2013.11928931. PMID 23543963
- [Background] Adams J, Berbarie RF. High-intensity cardiac rehabilitation training of a police officer for his return to work and sports after coronary artery bypass grafting. Proc (Bayl Univ Med Cent). 2013 Jan;26(1):39-41. doi: 10.1080/08998280.2013.11928911. PMID 23382610
- [Background] Adams J, Jordan S, Spencer K, Belanger J, Cheng D, Shock T, Karcher J. Energy expenditure in US automotive technicians and occupation-specific cardiac rehabilitation. Occup Med (Lond). 2013 Mar;63(2):103-8. doi: 10.1093/occmed/kqs192. Epub 2012 Nov 8. PMID 23144121
- [Background] Adams J, Hubbard M, McCullough-Shock T, Simms K, Cheng D, Hartman J, Strauss D, Anderson V, Lawrence A, Malorzo E. Myocardial work during endurance training and resistance training: a daily comparison, from workout session 1 through completion of cardiac rehabilitation. Proc (Bayl Univ Med Cent). 2010 Apr;23(2):126-9. doi: 10.1080/08998280.2010.11928599. PMID 20396420
- [Background] Adams J, Schneider J, Hubbard M, McCullough-Shock T, Cheng D, Simms K, Hartman J, Hinton P, Strauss D. Measurement of functional capacity requirements of police officers to aid in development of an occupation-specific cardiac rehabilitation training program. Proc (Bayl Univ Med Cent). 2010 Jan;23(1):7-10. doi: 10.1080/08998280.2010.11928571. PMID 20157495
- [Background] Adams J, Roberts J, Simms K, Cheng D, Hartman J, Bartlett C. Measurement of functional capacity requirements to aid in development of an occupation-specific rehabilitation training program to help firefighters with cardiac disease safely return to work. Am J Cardiol. 2009 Mar 15;103(6):762-5. doi: 10.1016/j.amjcard.2008.11.032. Epub 2009 Jan 24. PMID 19268728
- [Background] Naffe A, Iype M, Easo M, McLeroy SD, Pinaga K, Vish N, Wheelan K, Franklin J, Adams J. Appropriateness of sling immobilization to prevent lead displacement after pacemaker/implantable cardioverter-defibrillator implantation. Proc (Bayl Univ Med Cent). 2009 Jan;22(1):3-6. doi: 10.1080/08998280.2009.11928456. PMID 19169389
- [Background] Schmid J, Adams J, Cheng D. Cardiac rehabilitation of a 77-year-old male runner: consideration of the athlete, not the age. Proc (Bayl Univ Med Cent). 2009 Jan;22(1):16-8. doi: 10.1080/08998280.2009.11928460. PMID 19169393
- [Background] Adams J, Pullum G, Stafford P, Hanners N, Hartman J, Strauss D, Hubbard M, Lawrence A, Anderson V, McCullough T. Challenging traditional activity limits after coronary artery bypass graft surgery: a simulated lawn-mowing activity. J Cardiopulm Rehabil Prev. 2008 Mar-Apr;28(2):118-21. doi: 10.1097/01.HCR.0000314206.94428.9f. PMID 18360188
- [Background] Parker R, Adams JL, Ogola G, McBrayer D, Hubbard JM, McCullough TL, Hartman JM, Cleveland T. Current activity guidelines for CABG patients are too restrictive: comparison of the forces exerted on the median sternotomy during a cough vs. lifting activities combined with valsalva maneuver. Thorac Cardiovasc Surg. 2008 Jun;56(4):190-4. doi: 10.1055/s-2008-1038470. PMID 18481235
- [Background] Adams J, Cline M, Reed M, Masters A, Ehlke K, Hartman J. Importance of resistance training for patients after a cardiac event. Proc (Bayl Univ Med Cent). 2006 Jul;19(3):246-8. doi: 10.1080/08998280.2006.11928172. No abstract available. PMID 17252043
- [Background] Adams J, Cline MJ, Hubbard M, McCullough T, Hartman J. A new paradigm for post-cardiac event resistance exercise guidelines. Am J Cardiol. 2006 Jan 15;97(2):281-6. doi: 10.1016/j.amjcard.2005.08.035. Epub 2005 Nov 21. PMID 16442380

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-11): https://cdn.clinicaltrials.gov/large-docs/68/NCT05924568/Prot_SAP_000.pdf